CLINICAL TRIAL: NCT00874497
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Pilot Study to Assess the Pharmacodynamics, Efficacy and Safety of 50 mg Tetomilast Administered as Oral Tablets in Patients With Chronic Obstructive Pulmonary Disease Associated With Emphysema THIS STUDY IS CLOSED TO ENROLLMENT AND NEW SITES
Brief Title: Pilot Study of Tetomilast in Chronic Obstructive Pulmonary Disease (COPD) Associated With Emphysema
Acronym: EMPHASIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Terminated
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 197-08-250
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tetomilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 Tetomilast (Experimental)
  Interventions: Drug: tetomilast
- 2 Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tetomilast — Oral tetomilast 25 mg once daily for 2 weeks followed by 50 mg once daily for 2 years.
  Arms: 1 Tetomilast
Drug: placebo — Placebo for 104 weeks (2 years)
  Arms: 2 Placebo

SUMMARY:
Phase 2a multicenter, randomized, double-blind, placebo-controlled study to assess the pharmacodynamics, efficacy, and safety of tetomilast in patients with emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 40-75 yrs old,inclusive.
* Rating of greater than or equal to 1 on the Goddard scale in assessment of emphysema severity by HRCT.
* FEV1: FVC greater than 70% predicted.
* At least 1 documented COPD exacerbation within the past year but not within 8 weeks of randomization.
* Current or former smokers with a cigarette smoking history of at least 20 pack-years (or equivalent) and whose smoking status has not changed 60 days prior to screening.

Exclusion Criteria:

* Patients with asthma, active tuberculosis or bronchiectasis.
* A respiratory tract infection within 30 days prior to the screening visit.
* Any malignancy within the last 5 years with the exception of non-melanomatous skin cancer.
* Uncontrolled cardiovascular, endocrine, blood, or nervous system disorders.
* Uncontrolled condition with COPD exacerbation of level 2 or 3 in the 8-week period prior to randomization.
* Systemic use of corticosteroids or other immunosuppressive agents within 30 days of the screening visit.
* Subjects taking anticoagulants.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - UAB Lung Health Center, Birmingham, Alabama
  - Los Angeles Biomedical Institute, Torrance, California
  - Pulmonary Disease Specialist/PDS Research, Kissimmee, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Florida Premier Research Institute, Winter Park, Florida
  - Georgia Clinical Research, Austell, Georgia
  - Illinios Lung Institute, Peoria, Illinois
  - University of Louisville, Pulmonary Division, Louisville, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Texas Institute of Chest and Sleep Disorders, PA, Houston, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - Multicare Pulmonary Specialist, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 84 participants treated in the trial, 38 completed the trial and 10 participants were ongoing at the time the sponsor discontinued the trial.
Pre-assignment Details: Prior to randomization, each participant was in a 28- to 35-day screening period. Placebo was given for 14 days and a daily diary of symptom scores and actuations of albuterol/ipratropium bromide were collected.
Groups:
- Tetomilast 50 mg: Participants were administered oral tetomilast 25 milligram (mg) once daily for 2 weeks followed by 50 mg once daily for 102 weeks.
- Placebo: Participants were administered matching placebo for 104 weeks (2 years)
Period: Overall Study
Arm/Group | Tetomilast 50 mg | Placebo
Started | 51 (This is the number of participants who were treated and were considered as safety population.) | 33 (This is the number of participants who were treated and were considered as safety population.)
Completed | 23 | 15
Not Completed | 28 | 18
Not completed — Lost to Follow-up | 2 | 4
Not completed — Adverse Event | 9 | 4
Not completed — Sponsor Discontinued Trial | 7 | 3
Not completed — Met Withdrawal Criteria | 4 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized participants who had received study medication. Participants in this population were used for all demographic and safety summaries. Participants were analyzed based on the treatment which they had received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tetomilast 50 mg | Placebo | Total
Number analyzed (Participants) | 51 | 33 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (6.04) | 58.4 (7.71) | 58.2 (6.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 17 | 41
  Male | 27 | 16 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 104 in Trough Forced Expiratory Volume in 1 Second (FEV1)
Description: The analysis of the change from Baseline to Week 104 (last observation carried forward [LOCF]) in trough FEV1 is presented below.
Time Frame: Baseline to Week 104
Population: The Intent-to-Treat (ITT) population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable High-resolution computed tomography (HRCT) scan.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 48 | 28
L | -0.001 (0.2011) | -0.083 (0.3241)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis at Week 104; Test type: Superiority or Other; p = 0.1761, ANCOVA — P-values are based on Analysis of Covariance (ANCOVA) model of the change FEV1 from baseline to the specified study week using treatment group and current smoking status as fixed effects and the baseline FEV1 value as a covariate; Mean Difference (Final Values) = 0.0824, 95% CI 2-sided [-0.0378 to 0.2025]

2. Primary Outcome: Rate of Change From Baseline to Week 104 in 20th Percentile of Lung Density Voxels
Description: The analysis of the change from Baseline to Week 104 (LOCF) in the 20th percentile of lung density voxels (expressed in Hounsfield unit [HU] using quantitative HCRT) by visit and lung region is presented below.
Time Frame: Baseline to Week 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan. The number of participants analyzed at Week 104 were N = 43 and 25 respectively.
Measure: Mean (Standard Deviation); unit: Hounsfield unit/year
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 43 | 25
Hounsfield unit/year
  Right Upper (n= 43, 25) | -2.639 (7.9744) | 0.375 (7.1318)
  Right Middle (n= 43, 25) | -1.912 (6.0688) | -0.831 (7.1709)
  Right Lower (n= 43, 25) | -1.884 (11.5558) | 0.379 (11.0216)
  Left Upper (n= 43, 25) | -1.709 (9.8835) | 0.686 (8.0797)
  Left Lower (n= 43, 25) | -0.713 (11.3439) | 0.626 (11.4277)
  Right Whole (n= 43, 25) | -2.409 (7.3861) | -0.225 (7.7509)
  Left Whole (n= 43, 25) | -0.882 (9.8780) | 0.587 (8.9852)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Right Upper region of the lung at Week 104; Test type: Superiority or Other; p = 0.139, ANCOVA; Mean Difference (Final Values) = -2.904, 95% CI 2-sided [-6.77 to 0.97]
Statistical Analysis 2: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Right Middle region of the Lung at Week 104; Test type: Superiority or Other; p = 0.460, ANCOVA; Mean Difference (Final Values) = -1.210, 95% CI 2-sided [-4.46 to 2.04]
Statistical Analysis 3: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Right Lower region of the Lung at Week 104; Test type: Superiority or Other; p = 0.457, ANCOVA; Mean Difference (Final Values) = -2.176, 95% CI 2-sided [-7.98 to 3.63]
Statistical Analysis 4: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Left Upper region of the Lung at Week 104; Test type: Superiority or Other; p = 0.362, ANCOVA; Mean Difference (Final Values) = -2.167, 95% CI 2-sided [-6.88 to 2.54]
Statistical Analysis 5: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Left Lower region of the Lung at Week 104; Test type: Superiority or Other; p = 0.670, ANCOVA; Mean Difference (Final Values) = -1.225, 95% CI 2-sided [-6.94 to 4.48]
Statistical Analysis 6: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Right Whole region of the Lung at Week 104; Test type: Superiority or Other; p = 0.244, ANCOVA; Mean Difference (Final Values) = -2.218, 95% CI 2-sided [-5.98 to 1.55]
Statistical Analysis 7: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Left Whole region of the Lung at Week 104; Test type: Superiority or Other; p = 0.574, ANCOVA; Mean Difference (Final Values) = -1.374, 95% CI 2-sided [-6.23 to 3.48]

3. Secondary Outcome: Percent Change From Baseline in Trough FEV1 From Baseline to Week 104
Description: The percent change for the pulmonary function tests (PFT) from baseline was calculated for each study week as follows: % change from baseline = ([value at Week X - value at baseline] /value at baseline) x 100.
Time Frame: Baseline to Week 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan. The number of participants analyzed at Week 104 were N = 28 and 18 respectively.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 28 | 18
percentage change | -0.771 (14.4521) | -7.071 (22.9110)

4. Secondary Outcome: Density Mask Score Based on Specified Thresholds Including -950 HU
Description: The density mask score is defined as the percentage of lung density voxels that lie below a specified threshold in the lung region of interest. The higher the percentage of the participant's lung density voxels that lie below a specified threshold, the higher the level of the participant's emphysema in the lung region under consideration. Changes in the density mask score was assessed using only a single density mask threshold of -950 HU.
Time Frame: Baseline and Week 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan. The number of participants analyzed at Week 104 were N = 23 and 16 respectively.
Measure: Mean (Standard Deviation); unit: Hounsfield unit
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 23 | 16
Hounsfield unit
  Right Upper (n= 23, 16) | 0.57 (3.217) | -0.38 (4.425)
  Right Middle (n= 23, 16) | 0.96 (2.992) | -1.56 (4.980)
  Right Lower (n= 23, 16) | 1.17 (4.141) | -0.75 (4.494)
  Left Upper (n= 23, 16) | 1.17 (3.713) | -1.06 (4.823)
  Left Lower (n= 23, 16) | 1.22 (4.306) | -1.06 (5.221)
  Right Whole (n= 23, 16) | 0.96 (3.483) | -0.81 (4.151)
  Left Whole (n= 23, 16) | 1.09 (3.667) | -1.00 (4.719)
  Whole Lung (n= 23, 16) | 1.04 (3.431) | -1.00 (4.336)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Right Upper region of the Lung at Week 104; Test type: Superiority or Other; p = 0.436, ANCOVA; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [-1.53 to 3.47]
Statistical Analysis 2: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Right Middle region of the Lung at Week 104; Test type: Superiority or Other; p = 0.067, ANCOVA; Mean Difference (Final Values) = 2.31, 95% CI 2-sided [-0.17 to 4.79]
Statistical Analysis 3: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Right Lower region of the Lung at Week 104; Test type: Superiority or Other; p = 0.163, ANCOVA; Mean Difference (Final Values) = 1.97, 95% CI 2-sided [-0.83 to 4.77]
Statistical Analysis 4: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Left Upper region of the Lung at Week 104; Test type: Superiority or Other; p = 0.102, ANCOVA; Mean Difference (Final Values) = 2.27, 95% CI 2-sided [-0.48 to 5.02]
Statistical Analysis 5: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Left Lower region of the Lung at Week 104; Test type: Superiority or Other; p = 0.162, ANCOVA; Mean Difference (Final Values) = 2.11, 95% CI 2-sided [-0.89 to 5.12]
Statistical Analysis 6: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Right Whole region of the Lung at Week 104; Test type: Superiority or Other; p = 0.160, ANCOVA; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [-0.73 to 4.29]
Statistical Analysis 7: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Left Whole region of the Lung at Week 104; Test type: Superiority or Other; p = 0.122, ANCOVA; Mean Difference (Final Values) = 2.08, 95% CI 2-sided [-0.58 to 4.75]
Statistical Analysis 8: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of Whole Lung region of the Lung at Week 104; Test type: Superiority or Other; p = 0.106, ANCOVA; Mean Difference (Final Values) = 2.05, 95% CI 2-sided [-0.46 to 4.56]

5. Secondary Outcome: Rate of Change in the 20th Percentile of Lung Density Voxels Expressed in HU Units for the Whole Lung (Whole Right + Whole Left) From Baseline to Week 104
Description: The rate of change in lung density was calculated as the change in the 20th percentile of lung density voxels divided by the duration between the dates of measurement (month or year) where applicable. For example, if HRCT measurements are available over a span of 2 years, the annual rate of change was calculated as the difference over the 2 years divided by 2, where years between scans is given by years= floor(data of last scan - date of first scan + 1)/365.25.
Time Frame: Baseline to Week 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan. The number of participants analyzed at Week 104 were N = 46 and 26 respectively.
Measure: Mean (Standard Deviation); unit: Hounsfield unit/year
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 46 | 26
Hounsfield unit/year | -1.375 (7.909) | 0.115 (8.166)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; LS Mean Difference between Tetomilast and Placebo at Week 104; Test type: Superiority or Other; p = 0.469, ANCOVA; Mean Difference (Final Values) = -1.423, 95% CI 2-sided [-5.32 to 2.48]

6. Secondary Outcome: Observed Rate of Change in Emphysema From Baseline to Week 104
Description: The level of emphysema (g/L) within in a lung region is defined as the value of the selected percentile (10th, 15th, or 20th) in HU + 1000. The rate of change in the emphysema from baseline was calculated as the change in the level of emphysema from baseline to the specified visit divided by the time in years between the baseline and specified visit (i.e., [date of visit - date of baseline visit + 1]/365.25).
Time Frame: Baseline to Week 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 23 | 16
g/L
  Right Upper (n= 23, 16) | -0.64 (4.31) | 0.58 (6.27)
  Right Middle (n= 23, 16) | -0.87 (3.96) | 0.28 (5.77)
  Right Lower (n= 23, 16) | -0.53 (7.71) | 0.39 (9.16)
  Left Upper (n= 23, 16) | -1.49 (5.66) | 1.83 (7.04)
  Left Lower (n= 23, 16) | -0.62 (7.88) | 0.42 (9.62)
  Right Whole (n= 23, 16) | -0.79 (5.23) | 0.50 (6.78)
  Left Whole (n= 23, 16) | -0.95 (5.73) | 1.14 (7.73)
  Whole Lung (n= 23, 16) | -0.85 (5.30) | 0.74 (7.28)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right upper region of the lung at Week 104; Test type: Superiority or Other; p = 0.519, ANCOVA; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-4.42 to 2.27]
Statistical Analysis 2: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right middle region of the lung at Week 104; Test type: Superiority or Other; p = 0.463, ANCOVA; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-3.92 to 1.82]
Statistical Analysis 3: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right lower region of the lung at Week 104; Test type: Superiority or Other; p = 0.598, ANCOVA; Mean Difference (Final Values) = -1.40, 95% CI 2-sided [-6.74 to 3.94]
Statistical Analysis 4: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left upper region of the lung at Week 104; Test type: Superiority or Other; p = 0.142, ANCOVA; Mean Difference (Final Values) = -2.94, 95% CI 2-sided [-6.92 to 1.03]
Statistical Analysis 5: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left lower region of the lung at Week 104; Test type: Superiority or Other; p = 0.757, ANCOVA; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-6.26 to 4.59]
Statistical Analysis 6: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right whole region of the lung at Week 104; Test type: Superiority or Other; p = 0.500, ANCOVA; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-5.03 to 2.50]
Statistical Analysis 7: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left whole region of the lung at Week 104; Test type: Superiority or Other; p = 0.353, ANCOVA; Mean Difference (Final Values) = -1.93, 95% CI 2-sided [-6.09 to 2.23]
Statistical Analysis 8: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of whole region of the lung at Week 104; Test type: Superiority or Other; p = 0.438, ANCOVA; Mean Difference (Final Values) = -1.52, 95% CI 2-sided [-5.43 to 2.40]

7. Secondary Outcome: Change From Baseline to Week 104 in Cumulative Frequency of HU
Description: The area under the curve (AUC) is defined as the cumulative voxel frequency in HU (ie, the value of the density mask denominator). Blood samples (4 mL) for pharmacokinetic analysis were collected for the determination of plasma OPC-6535 concentrations at Predose on Day 1 and Weeks 26, 52, 78 and 104.
Time Frame: Baseline and Week 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hounsfield unit*hour
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 23 | 16
Hounsfield unit*hour
  Right Upper (n= 23, 16) | 4429363 (1696731) | 4596228 (1012400)
  Right Middle (n= 23, 16) | 1474625 (409858) | 1500073 (644286)
  Right Lower (n= 23, 16) | 4507375 (1302992) | 4498652 (1703957)
  Left Upper (n= 23, 16) | 4818524 (1541192) | 5105606 (1574676)
  Left Lower (n= 23, 16) | 4351407 (1677740) | 4392819 (1256283)
  Right Whole (n= 23, 16) | 10411363 (2651975) | 10594953 (2678348)
  Left Whole (n= 23, 16) | 9169931 (2630471) | 9498425 (2471947)
  Whole Lung (n= 23, 16) | 19581293 (5212292) | 20093377 (5022730)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right upper region of the lung at Week 104; Test type: Superiority or Other; p = 0.220, ANCOVA; Mean Difference (Final Values) = 351487, 95% CI 2-sided [-219976 to 922951]
Statistical Analysis 2: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right middle region of the lung at Week 104; Test type: Superiority or Other; p = 0.146, ANCOVA; Mean Difference (Final Values) = 103036, 95% CI 2-sided [-37651 to 243723]
Statistical Analysis 3: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right lower region of the lung at Week 104; Test type: Superiority or Other; p = 0.322, ANCOVA; Mean Difference (Final Values) = 247358, 95% CI 2-sided [-252728 to 747444]
Statistical Analysis 4: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left upper region of the lung at Week 104; Test type: Superiority or Other; p = 0.141, ANCOVA; Mean Difference (Final Values) = 362384, 95% CI 2-sided [-126518 to 851286]
Statistical Analysis 5: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left lower region of the lung at Week 104; Test type: Superiority or Other; p = 0.325, ANCOVA; Mean Difference (Final Values) = 294202, 95% CI 2-sided [-303329 to 891733]
Statistical Analysis 6: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right whole region of the lung at Week 104; Test type: Superiority or Other; p = 0.258, ANCOVA; Mean Difference (Final Values) = 575882, 95% CI 2-sided [-439692 to 1591457]
Statistical Analysis 7: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left whole region of the lung at Week 104; Test type: Superiority or Other; p = 0.247, ANCOVA; Mean Difference (Final Values) = 589373, 95% CI 2-sided [-426928 to 1605673]
Statistical Analysis 8: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of whole lung region of the lung at Week 104; Test type: Superiority or Other; p = 0.251, ANCOVA; Mean Difference (Final Values) = 1156318, 95% CI 2-sided [-855009 to 3167645]

8. Secondary Outcome: Change From Baseline to Week 104 in Computed Tomography (CT) - Derived Lung Volumes (Total Lung Capacity [TLC] and Residual Volume [RV])
Description: Change from baseline in CT-derived lung volumes TLC and RV are presented in the below outcome data table.
Time Frame: Baseline to Week 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan. The number of participants analyzed at Week 104 were N = 22 and 16 respectively.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 22 | 16
mL
  Right Upper (RV) (n= 22, 16) | 31.4 (145.3) | -64.3 (216.5)
  Right Middle (RV) (n= 22, 16) | -14.1 (65.7) | -8.6 (63.6)
  Right Lower (RV) (n= 22, 16) | 18.1 (186.2) | -49.3 (254.8)
  Left Upper (RV) (n= 22, 16) | 11.0 (153.8) | -72.9 (212.9)
  Left Lower (RV) (n= 22, 16) | 13.0 (216.2) | -52.8 (220.7)
  Right Whole (RV) (n= 22, 16) | 35.3 (350.7) | -122.1 (504.5)
  Left Whole (RV) (n= 22, 16) | 23.8 (352.0) | -125.6 (401.8)
  Whole Lung (RV) (n= 22, 16) | 59.4 (693.3) | -247.8 (894.2)
  Right Upper (TLC) (n= 22, 16) | -0.7 (173.9) | -52.3 (144.5)
  Right Middle (TLC) (n= 22, 16) | 3.7 (71.2) | -6.1 (62.6)
  Right Lower (TLC) (n= 22, 16) | -12.5 (215.2) | -18.1 (159.2)
  Left Upper (TLC) (n= 22, 16) | 1.0 (141.8) | -59.1 (139.2)
  Left Lower (TLC) (n= 22, 16) | -6.9 (270.2) | -35.8 (195.6)
  Right Whole (TLC) (n= 22, 16) | -9.2 (341.0) | -76.3 (291.0)
  Left Whole (TLC) (n= 22, 16) | -6.1 (390.6) | -95.1 (320.9)
  Whole Lung (TLC) (n= 22, 16) | -15.2 (711.3) | -171.4 (584.4)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right upper lung region (RV) at Week 104; Test type: Superiority or Other; p = 0.181, ANCOVA; Mean Difference (Final Values) = 77.9, 95% CI 2-sided [-38.0 to 193.8]
Statistical Analysis 2: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right middle lung region (RV) at Week 104; Test type: Superiority or Other; p = 0.781, ANCOVA; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-48.8 to 36.9]
Statistical Analysis 3: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right lower lung region (RV) at Week 104; Test type: Superiority or Other; p = 0.445, ANCOVA; Mean Difference (Final Values) = 47.7, 95% CI 2-sided [-77.8 to 173.2]
Statistical Analysis 4: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left upper lung region (RV) at Week 104; Test type: Superiority or Other; p = 0.259, ANCOVA; Mean Difference (Final Values) = 62.6, 95% CI 2-sided [-48.1 to 173.2]
Statistical Analysis 5: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left lower lung region (RV) at Week 104; Test type: Superiority or Other; p = 0.639, ANCOVA; Mean Difference (Final Values) = 32.0, 95% CI 2-sided [-105.6 to 169.6]
Statistical Analysis 6: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right whole lung region (RV) at Week 104; Test type: Superiority or Other; p = 0.408, ANCOVA; Mean Difference (Final Values) = 102.3, 95% CI 2-sided [-145.9 to 350.5]
Statistical Analysis 7: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left whole lung region (RV) at Week 104; Test type: Superiority or Other; p = 0.445, ANCOVA; Mean Difference (Final Values) = 85.2, 95% CI 2-sided [-138.8 to 309.2]
Statistical Analysis 8: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of whole lung region (RV) at Week 104; Test type: Superiority or Other; p = 0.421, ANCOVA; Mean Difference (Final Values) = 187.6, 95% CI 2-sided [-279.6 to 654.8]
Statistical Analysis 9: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right upper lung region (TLC) at Week 104; Test type: Superiority or Other; p = 0.353, ANCOVA; Mean Difference (Final Values) = 50.7, 95% CI 2-sided [-58.5 to 159.9]
Statistical Analysis 10: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right middle lung region (TLC) at Week 104; Test type: Superiority or Other; p = 0.660, ANCOVA; Mean Difference (Final Values) = 9.9, 95% CI 2-sided [-35.3 to 55.0]
Statistical Analysis 11: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right lower lung region (TLC) at Week 104; Test type: Superiority or Other; p = 0.859, ANCOVA; Mean Difference (Final Values) = 10.7, 95% CI 2-sided [-110.7 to 132.1]
Statistical Analysis 12: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left upper lung region (TLC)at Week 104; Test type: Superiority or Other; p = 0.253, ANCOVA; Mean Difference (Final Values) = 51.5, 95% CI 2-sided [-38.4 to 141.4]
Statistical Analysis 13: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left lower lung region (TLC) at Week 104; Test type: Superiority or Other; p = 0.754, ANCOVA; Mean Difference (Final Values) = 23.3, 95% CI 2-sided [-126.0 to 172.6]
Statistical Analysis 14: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of right whole lung region (TLC) at Week 104; Test type: Superiority or Other; p = 0.546, ANCOVA; Mean Difference (Final Values) = 62.2, 95% CI 2-sided [-145.1 to 269.5]
Statistical Analysis 15: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of left whole lung region (TLC) at Week 104; Test type: Superiority or Other; p = 0.554, ANCOVA; Mean Difference (Final Values) = 64.9, 95% CI 2-sided [-155.5 to 285.3]
Statistical Analysis 16: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis of whole lung region (TLC) at Week 104; Test type: Superiority or Other; p = 0.524, ANCOVA; Mean Difference (Final Values) = 132.2, 95% CI 2-sided [-284.9 to 549.4]

9. Secondary Outcome: Change From Baseline to Week 104 in Trough RV/TLC
Description: Change from Baseline in Trough RV/TLC is presented in the below outcome data table.
Time Frame: Baseline to Week 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan. The number of participants analyzed at Week 104 were n= 21 and 14 respectively.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 21 | 14
unitless | 0.01 (0.12) | 0.01 (0.07)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Test type: Superiority or Other; p = 0.5843, ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.07 to 0.04]

10. Secondary Outcome: Change From Baseline to Week 104 in Trough Inspiratory Capacity
Description: Change from Baseline in Trough Inspiratory Capacity is presented in the below outcome data table.
Time Frame: Baseline toWeek 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan. The number of participants analyzed at Week 104 were N = 25 and 14 respectively.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 25 | 14
mL | 0.074 (0.574) | -0.225 (0.384)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Test type: Superiority or Other; p = 0.1252, ANCOVA; Mean Difference (Final Values) = 0.249, 95% CI 2-sided [-0.073 to 0.571]

11. Secondary Outcome: Change From Baseline to Week 104 in Trough Functional Residual Capacity (FRCpleth)
Description: Change from baseline in trough FRCpleth is presented in the below outcome data table.
Time Frame: Baseline to Week 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan. The number of participants analyzed at Week 104 were N = 23 and 15 respectively.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 23 | 15
mL | -0.010 (1.0130) | 0.029 (0.5290)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Test type: Superiority or Other; p = 0.4661, ANCOVA; Mean Difference (Final Values) = -0.1835, 95% CI 2-sided [-0.6892 to 0.3221]

12. Secondary Outcome: Change From Baseline to Week 104 in Carbon Monoxide Diffusion Capacity (DLco)
Description: Change from Baseline in DLco is presented in the below outcome data table.
Time Frame: Baseline to Week 104
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmoL/min/kPA
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 23 | 15
mmoL/min/kPA | 0.021 (0.8485) | -0.625 (1.6288)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Test type: Superiority or Other; p = 0.134, ANCOVA; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-0.19 to 1.40]

13. Secondary Outcome: Change From Baseline to Week 104 in Mean Specific Airway Resistance (sRaw) and Specific Conductance (sGaw)
Description: Change from baseline in sRaw and sGaw is presented in the below outcome data table.
Time Frame: Baseline to Week 104
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: kPa.sec
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 23 | 15
kPa.sec
  sRaw | -0.29 (1.110) | 0.47 (1.387)
  sGaw | 0.11 (0.584) | -0.07 (0.293)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis for sRaw; Test type: Superiority or Other; p = 0.074, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.50 to 0.07]
Statistical Analysis 2: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis for sGaw; Test type: Superiority or Other; p = 0.155, ANCOVA; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.09 to 0.52]

14. Secondary Outcome: Change From Baseline to Week 104 in 7-day Average Total Symptom Score of Dyspnea, Cough and Sputum
Description: Participants used the Breathlessness, Cough, and Sputum Scale (BCSS) as the diary to daily monitor and rate their symptoms of difficulty breathing, cough, and sputum. The scale allows patients to rate each symptom on a scale of 0 (no difficultly for breathing and sputum, or unaware of coughing) to 4 (an almost constant problem for breathing and sputum, or almost constant for cough).
Time Frame: Baseline to Week 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan. The number of participants analyzed at Week 104 were N = 13 and 9 respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 13 | 9
units on a scale
  Mean prior daily breath symptoms (n= 13, 9) | 0.13 (0.60) | 0.20 (0.95)
  Mean prior daily cough symptoms (n= 13, 9) | 0.10 (0.40) | -0.13 (1.13)
  Mean prior daily sputum symptoms (n= 13, 9) | 0.15 (0.74) | 0.31 (1.07)
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis for mean prior daily breath symptoms; Test type: Superiority or Other; p = 0.845, ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.77 to 0.64]
Statistical Analysis 2: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis for mean prior daily cough symptoms; Test type: Superiority or Other; p = 0.549, ANCOVA; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.52 to 0.94]
Statistical Analysis 3: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis for mean prior daily sputum symptoms; Test type: Superiority or Other; p = 0.717, ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.93 to 0.65]

15. Secondary Outcome: Change From Baseline to Week 104 in 7-day Mean Number of Actuations of Rescue Medications
Description: Participants recorded rescue medication use (albuterol and/or ipratropium bromide) in a rescue medication log.
Time Frame: Baseline to Week 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan. The number of participants analyzed at Week 104 were N = 14 and 9 respectively.
Measure: Mean (Standard Deviation); unit: number of puffs
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 14 | 9
number of puffs | -0.74 (1.57) | -2.52 (3.82)

16. Secondary Outcome: Percentage of Participants With COPD Exacerbations by Group at Week 104
Description: For the COPD exacerbations, baseline is defined as Randomization (Day 1). COPD exacerbations, defined as an acute worsening of COPD symptoms, were classified as being in one of 3 levels: Level I (can by self-managed by the participant); Level II (requires a physician visit), or Level III (requires a hospital visit).
Time Frame: Baseline and Week 104
Population: The ITT population consisted of all randomized participants with non-missing baseline data and at least one post-baseline trough FEV1 measurement or evaluable HRCT scan.
Measure: Number; unit: percentage of participants
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 48 | 28
percentage of participants
  Level I (Baseline) (n= 48, 28) | 0.0 | 0.0
  Level I (Week 104) (n= 23, 15) | 4.3 | 6.7
  Level II (Baseline) (n= 48, 28) | 0.0 | 0.0
  Level II (Week 104) (n= 23, 15) | 8.7 | 6.7
  Level III (Baseline) (n= 48, 28) | 0.0 | 0.0
  Level III (Week 104) (n= 23, 15) | 8.7 | 0.0
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis for level I (self management) at week 104; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis for level II (physician visit) at week 104; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis for level III (hospital visit) at week 104; Test type: Superiority or Other; p = 0.5092, Fisher Exact

17. Secondary Outcome: Percentage of Participants Experiencing a COPD Exacerbation (Level 2 or Higher)
Description: Percentage of participants experiencing a COPD exacerbation in a level 2 or higher are presented in the below outcome data table.
Time Frame: Baseline and Week 104
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Tetomilast 50 mg | Placebo
Number analyzed (Participants) | 48 | 28
percentage of participants
  Level 2 or Higher (Baseline) | 0.0 | 0.0
  Level 1 or No Exacerbation (Baseline) | 100.0 | 100.0
  Level 2 or Higher (Week 104) | 8.3 | 3.6
  Level 1 or No Exacerbation (Week 104) | 39.6 | 50.0
Statistical Analysis 1: Comparison: Tetomilast 50 mg vs Placebo; Statistical analysis at Week 104; Test type: Superiority or Other; p = 0.630, Fisher Exact — Fisher's Exact test was used to determine whether the tetomilast and placebo groups differ in the proportion of participants who experienced Level 2 or higher COPD exacerbations during the study

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent, throughout the 104 week treatment period until the follow-up visit of 14 (+2) days.
Groups:
- Tetomilast 25 mg: Participants were administered oral tetomilast 25 milligram (mg) once daily for 2 weeks followed by 50 mg once daily for 102 weeks.
Arm/Group | Tetomilast 25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 13/51 | 12/33
Other Adverse Events (participants affected / at risk) | 30/51 | 23/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tetomilast 25 mg (N=51) | Placebo (N=33)
Pneumonia (Infections and infestations) | 2 | 3
Lobar Pneumonia (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Colostomy infection (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Chronic obstrutive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tetomilast 25 mg (N=51) | Placebo (N=33)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Gastritis (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Pyrexia (General disorders) | 0 | 2
Bronchitis (Infections and infestations) | 5 | 6
Gastroenteritis viral (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Urinary tract infection (Infections and infestations) | 3 | 3
Weight decreased (Investigations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 2 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 0
Chronic obstrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 3 | 2

LIMITATIONS AND CAVEATS:
This trial was terminated early, not due to a safety concern, but due to a business decision to cease development of the tetolimast clinical program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.